CLINICAL TRIAL: NCT04037787
Title: ERAS (Enhanced Recovery After Surgery) Protocol Implementation in Piedmont Region for Colorectal Cancer Surgery. A Stepped-wedge Cluster Randomized Clinical Trial
Brief Title: ERAS (Enhanced Recovery After Surgery) Protocol Implementation in Piedmont Region for Colorectal Cancer Surgery
Acronym: ERAS-Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other); Ministry of Health, Italy (Other Government); Regione Piemonte (Other)
Responsible Party: Principal Investigator, Felice Borghi, Surgeon, Ospedale Santa Croce-Carle Cuneo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ERAS-Colon-Piemonte
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Quality Improvement; Perioperative Care; Recovery of Function
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Enhanced Recovery After Surgery; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized clinical trial. Each center starts as control group (usual care) and switch to experimental group (ERAS protocol implementation) according to a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Perioperative care for colorectal cancer cancer is managed according to current hospital clinical practice.
- ERAS protocol (Experimental): Perioperative care for colorectal cancer surgery is managed according to ERAS protocol.
  Interventions: Procedure: ERAS protocol

INTERVENTIONS:
Procedure: ERAS protocol — In colorectal cancer surgery, the ERAS protocol involves an accurate interview with the patient in the preoperative phase aimed at smoking and alcohol cessation, the reduction of preoperative fasting with administration of oral carbohydrates before surgery, use of intestinal preparation for selected cases only (rectal surgery), the prophylaxis of thromboembolism, a correct antibiotic prophylaxis, the prevention of intraoperative hypothermia, prevention of volume overload, preference for minimally invasive surgery, prevention of postoperative nausea and vomiting, very limited use of the nasogastric tube, early removal of the urinary catheter, multimodal analgesia to minimize opiate consumption, early postoperative mobilization and early post-operative feeding, to promote rapid recovery of gastro-intestinal functions.
  Other Names: ERAS (Enhanced Recovery After Surgery) protocol
  Arms: ERAS protocol

SUMMARY:
The study assesses the impact on quality of care of implementing the ERAS (Enhanced Recovery After Surgery) protocol for colorectal cancer surgery in the network of public hospitals in the Regione Piemonte (North-West Italy). Every hospital is a cluster entering the study treating patients according to its current clinical practice. On the basis of a randomized order, each hospital switches from current clinical practice to the adoption of the ERAS protocol.

DETAILED DESCRIPTION:
ERAS (Enhanced Recovery After Surgery) protocol is a multimodal perioperative care pathways designed to achieve early recovery after surgical procedures by maintaining preoperative organ function and reducing the profound stress response following surgery. Even if efficacy and safety of ERAS protocol in colorectal surgery is well-established in the literature, its implementation is limited to few selected centres in Piemonte. The aim of the study is to extend the implementation of the ERAS protocol to whole regional network of hospitals. Specific objectives are to estimate its impact on different dimensions of quality of care, including length of stay, complications and patient satisfaction, and to identify possible barriers or facilitating factors.

ELIGIBILITY:
Inclusion Criteria:

* All the hospital wards within the Piemonte Region performing colorectal cancer surgery
* All the patients receiving an elective surgery for colorectal cancer, with or without protective stoma.

Exclusion Criteria:

* Hospital wards performing less than 30 expected cases per year
* Emergency surgery
* High severity cases not allowing ERAS protocol implementation (i.e. American Society of Anesthesiologists score: ASA V).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2397 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Length of stay | 22 days after admission
  Mean length of stay calculated as difference between date of discharge and date of admission of the hospitalization for surgery, excluding length of stay >94th percentile of the expected distribution (expected 22 days).

SECONDARY OUTCOMES:
Length of stay >22 days | 30 days after admission
  Rate of patients with a length of stay >22 days
Recovery after surgery | 24 hours after surgery
  Score of quality of recovery at 24 hours after surgery, assessed with the questionnaire Quality of Recovery (QoR-15), a 15-items instrument, with responses recorded on a 11-point Likert-type scale form 0 (worst scenario) to 10 (best scenario) and an overall score ranging from 0 (poor recovey) to 150 (excellent recovery).
  A visual analogue scale (VAS), ranging from 0 (worst imaginable health state) to 10 (worst imaginable health state) is also supplied as summary evaluation.
Complications | 30 days after discharge
  Rate of surgical and medical complication after surgery For surgical complications: Comprehensive Complication Index
Transfer to intensive care unit | 30 days after surgery
  Rate of transfers to intensive care unit after surgery
Emergency visits after discharge | 30 days after discharge
  Rate of emergency visit in the first month after discharge
Hospital admissions after discharge | 30 days after discharge
  Rate of new admissions in the first month after discharge
Reintervention | 30 days after surgery
  Rate of reintervention in the first month after surgery, excluding planned interventions
Patients' satisfaction | 15 days after discharge
  Score of patients' satisfaction measured 2 weeks after discharge, assessed with the questionnaire Surgical Satisfaction Questionnaire (SSQ8) supplied by telephone. SSQ8 is a 8-items instrument, with responses recorded on a 5-point Likert-type scale from 0 (worst scenario) to 4 (best scenario) and an overall score ranging from 0 (very unsatisfied) to 32 (very satisfied).
Healthcare costs | 30 days after discharge
  Mean healthcare costs from pre admission visit to 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Giovannino Ciccone, MD, Study Chair — Azienda Ospedaliera Universitaria Città della Salute e della Scienza di Torino
Locations (1):
- Ospedale Santa Croce-Carle Cuneo, Cuneo, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be made available upon reasonable request, with appropriate human research ethics approvals and data transfer agreements in place.
Supporting Information: Study Protocol
Time Frame: Available after results publication
Access Criteria: Upon reasonable request, with appropriate human research ethics approvals and data transfer agreements in place.

REFERENCES:
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Kehlet H. Fast-track surgery-an update on physiological care principles to enhance recovery. Langenbecks Arch Surg. 2011 Jun;396(5):585-90. doi: 10.1007/s00423-011-0790-y. Epub 2011 Apr 6. PMID 21468643
- [Background] Greco M, Capretti G, Beretta L, Gemma M, Pecorelli N, Braga M. Enhanced recovery program in colorectal surgery: a meta-analysis of randomized controlled trials. World J Surg. 2014 Jun;38(6):1531-41. doi: 10.1007/s00268-013-2416-8. PMID 24368573
- [Background] Braga M, Borghi F, Scatizzi M, Missana G, Guicciardi MA, Bona S, Ficari F, Maspero M, Pecorelli N; PeriOperative Italian Society. Impact of laparoscopy on adherence to an enhanced recovery pathway and readiness for discharge in elective colorectal surgery: Results from the PeriOperative Italian Society registry. Surg Endosc. 2017 Nov;31(11):4393-4399. doi: 10.1007/s00464-017-5486-0. Epub 2017 Mar 13. PMID 28289972
- [Background] Greer NL, Gunnar WP, Dahm P, Lee AE, MacDonald R, Shaukat A, Sultan S, Wilt TJ. Enhanced Recovery Protocols for Adults Undergoing Colorectal Surgery: A Systematic Review and Meta-analysis. Dis Colon Rectum. 2018 Sep;61(9):1108-1118. doi: 10.1097/DCR.0000000000001160. PMID 30086061
- [Derived] Pagano E, Pellegrino L, Robella M, Castiglione A, Brunetti F, Giacometti L, Rolfo M, Rizzo A, Palmisano S, Meineri M, Bachini I, Morino M, Allaix ME, Mellano A, Massucco P, Bellomo P, Polastri R, Ciccone G, Borghi F; ERAS-colorectal Piemonte group. Implementation of an enhanced recovery after surgery protocol for colorectal cancer in a regional hospital network supported by audit and feedback: a stepped wedge, cluster randomised trial. BMJ Qual Saf. 2024 May 17;33(6):363-374. doi: 10.1136/bmjqs-2023-016594. PMID 38423752
- [Derived] Pagano E, Pellegrino L, Rinaldi F, Palazzo V, Donati D, Meineri M, Palmisano S, Rolfo M, Bachini I, Bertetto O, Borghi F, Ciccone G; ERAS Colon-Rectum Piemonte study group members. Implementation of the ERAS (Enhanced Recovery After Surgery) protocol for colorectal cancer surgery in the Piemonte Region with an Audit and Feedback approach: study protocol for a stepped wedge cluster randomised trial: a study of the EASY-NET project. BMJ Open. 2021 Jun 3;11(6):e047491. doi: 10.1136/bmjopen-2020-047491. PMID 34083345